CLINICAL TRIAL: NCT06042569
Title: Dose Reduction of Docetaxel-Based Chemotherapy in Vulnerable Older Women With Early-Stage Breast Cancer (DOROTHY)
Brief Title: Dose-Reduced Docetaxel With Cyclophosphamide for the Treatment of Vulnerable Older Women With Stage I-III HER2 Negative Breast Cancer, the DOROTHY Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rising Tide Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21374; NCI-2023-06506 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21374 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-09-07; First posted 2023-09-18 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; HER2-Negative Breast Carcinoma
MeSH Terms: interventions — Cyclophosphamide; Docetaxel

STUDY DESIGN:
Masking Description: Randomization module also conceals allocation from other study personnel except the biostatistician and the designated study coordinator by limiting their user's right.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I: (Dose-reduced docetaxel, cyclophosphamide) (Experimental): Patients receive dose-reduced docetaxel IV over 60 minutes and cyclophosphamide IV over 30 minutes on day 1 of each cycle. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Docetaxel; Other: Medical Chart Review; Other: Questionnaire Administration
- Arm II: (Standard dose docetaxel, cyclophosphamide) (Active Comparator): Patients receive standard dose docetaxel IV over 60 minutes and cyclophosphamide IV over 30 minutes on day 1 of each cycle. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Docetaxel; Other: Medical Chart Review; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Other: Medical Chart Review — Ancillary studies
  Other Names: Chart Review
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests how well dose-reduced docetaxel combined with cyclophosphamide works in treating older women with early stage (stage I-III) HER2 negative breast cancer vulnerable to toxicity. Chemotherapy drugs, such as docetaxel and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Docetaxel and cyclophosphamide are commonly used, but is not well tolerated at the standard dose and can affect the way older patients feel physically and emotionally. Giving dose-reduced docetaxel combined with cyclophosphamide may be an effective treatment option and improve quality of life in vulnerable older women with stage I-III HER2 negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Compare the relative dose intensity (RDI) of reduced- versus (vs.) standard-dose docetaxel dosing strategies.

SECONDARY OBJECTIVE:

I. Compare treatment tolerability of reduced- vs. standard-dose docetaxel dosing strategies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive dose-reduced docetaxel intravenously (IV) over 60 minutes and cyclophosphamide IV over 30 minutes on day 1 of each cycle. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive standard dose docetaxel IV over 60 minutes and cyclophosphamide IV over 30 minutes on day 1 of each cycle. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days then at least twice yearly for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provided informed consent or a legally authorized representative is able to consent on behalf of the patient
* Willing to answer questionnaires as part of their participation
* Age: >= 65 years by the time of study registration
* Histologically or cytologically confirmed breast cancer(s) that is human epidermal growth factor receptor 2 negative (HER2-negative) per the most recent 2018 American Society of Clinical Oncology College of American Pathologists (ASCO CAP) guidelines relapsed/ refractory disease
* Estrogen receptor and progesterone receptor immunohistochemistry (IHC) status must be known; any estrogen receptor (ER)/progesterone receptor (PR) status is eligible
* Non-metastatic, invasive breast cancer (scans are not required to document non-metastatic disease- any staging work-up is up to the treating providers' discretion)
* Recommended to have either standard dose neoadjuvant docetaxel, cyclophosphamide (TC) chemotherapy or adjuvant TC chemotherapy per their treating provider. Participant may be on immunotherapy concurrently with the protocol regimen at the discretion of the treating physician
* Any surgery, nodal assessment, radiation, hormonal therapy is left up to the treating provider but should not occur concurrently with study therapy
* Any patient who received pre-operative hormonal therapy and who is then recommended for neo/adjuvant chemotherapy is eligible, though hormonal therapy should be held during study treatment administration
* For patients with bilateral or multifocal/multicentric breast cancers, the following criteria must be met to enroll: (1) both cancer are HER2 negative, AND (2) the provider feels the patient will benefit from TC for at least one of the cancers
* Patients who do not speak or read English are eligible as long as adequate interpreter services are available or the surveys are available in the preferred language (i.e. the Geriatric Assessment [GA] and Patient Reported Outcomes [PRO] surveys are available in many languages)

Exclusion Criteria:

* Participants who have already received any chemotherapy for their current breast cancer
* Patients with recurrent and/or metastatic disease will be excluded. Prior diagnoses of breast cancers (including ductal carcinoma in situ [DCIS]) are allowed, provided that the treating provider feels that the current cancer most likely represents a new primary breast cancer and not recurrent disease
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cyclophosphamide and/or docetaxel
* Past treatment with the regimen TC for prior breast cancer

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2030-03-20 (Estimated); Study Completion 2030-03-20 (Estimated)

PRIMARY OUTCOMES:
Relative dose intensity (RDI) | At completion of 4 cycles, up to 12 weeks (each cycle is every three weeks)
  RDI is defined as the ratio of actual dose intensity received to the standard dose intensity, ranging from 0 to 100%. The RDI between the two arms will be compared using T-test, RDI difference and 90% confidence interval. A one-sided p-value < 0.05 will be considered statistically significant.

SECONDARY OUTCOMES:
Treatment success | At completion of 4 cycles, up to 12 weeks (Each cycle is three weeks)
  Treatment success is defined as the proportion of patients who receive all 4 planned cycles of chemotherapy without unacceptable toxicity (grade 3-4), hospitalization/death at the end of treatment, and without decline in physical function status. Proportion of treatment success between the 2 arms will be compared using Chi-square test. A one-sided p-value of < 0.05 will be considered statistically significant.
Patient-reported symptomatic toxicities | At each chemotherapy cycle for 4 cycles, end of treatment and at 3, 6, 12 and 24 months after treatment ends)(Each cycle is three weeks).
  Toxicities will be described using the National Cancer Institute (NCI) Patient Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE). Patient reported outcomes will evaluate how well symptoms reported correlate/agree with clinician reported adverse events.
Differences in PRO-CTCAE and clinician-reported toxicities | At each chemotherapy cycle for 4 cycles and at 3, 6, 12, and 24 months after treatment ends (Each cycle is three weeks).
  Treatment related toxicities grade 3 or higher experienced by patients between the 2 arms will be described using NCI-CTCAE version (v) 5.0. Chi-square or Fisher exact test will be used to explore the difference in terms of rate of PRO-CTCAE and clinician reported CTCAE between the 2 arms at the end of chemotherapy. Agreement proportions between PRO-CTCAE and clinician reported CTCAE will be explored and calculated for the 2 arms combined.
Patient satisfaction | Up to 3 months after treatment ends
  Patient-reported satisfaction will be measured using the Was It Worth It questionnaire. Data will be scored and summarized according to their scoring manual. Chi-square or Fisher exact test will be used to compare the proportion of patients who consider it worthwhile to undergo treatment, the proportion of patients who would undergo the treatment again, and the proportionof patients who would recommend the treatment to others between the 2 arms.
Changes in function and health status | At baseline and at 3, 6, 12 and 24 months after treatment ends
  Elements of the Geriatric Assessment (GA) will be used to calculate the deficit accumulation index for each patient on each study arm over time. Trajectories of change in function will be examined. Data will be scored and summarized according to the GA scoring manual.
Incidence of adverse events | At every 3 weeks up to completion of study treatment
  Toxicity experienced by patients for each arm at each cycle will be described using NCI CTCAE v 5.0. Hematologic and non-hematologic toxicities will be examined by grade, type and offending agent.
Invasive disease-free survival | Up to 2 years
  Defined as an occurrence of ipsilateral invasive breast cancer recurrence, regional invasive breast cancer recurrence, distant recurrence, death attributable to any cause, contralateral invasive breast cancer and second non-breast invasive cancer.
Local recurrences | Up to 3 years
  Local recurrence will be defined as the number of in-breast, chest wall after mastectomy and axillary recurrences.
Distant recurrences | Up to 2 years
  Distant recurrence will be defined as the number of recurrences occurring with or without localized recurrence that have occurred distant to the breast.
Overall survival | From registration to death due to any cause up to 24 months
  Breast cancer-specific survival and cause of death will also be examined.
Progression-free survival | From registration to the earliest of progression or death due to any cause up to 24 months
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse. In a clinical trial, measuring the progression-free survival is one way to see how well a new treatment works.

CONTACTS AND LOCATIONS:
Overall Officials: Thanh Nga E Doan, MD, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts